CLINICAL TRIAL: NCT04443114
Title: Assessing the Feasibility of Peer-Led Educational Workshops on Increasing Awareness Among American Muslims About Living Donation in Mosque Communities
Brief Title: Informing American Muslims About Living Donation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB18-1378
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Living Organ Donation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Arm (Other): The early arm will receive the experimental organ donation workshop first, followed by the control workshop on end-of-life care.
  Interventions: Other: Organ Donation Workshop; Other: End of Life Care Workshop
- Late Arm (Other): The late arm will receive the control workshop on end-of-life care first, followed by the experimental organ donation workshop.
  Interventions: Other: Organ Donation Workshop; Other: End of Life Care Workshop

INTERVENTIONS:
Other: Organ Donation Workshop — Discussion Moderated by Peer Educators Didactic Session 1: Biomedical Aspects of Living Donation Didactic Session 2: Organ Donation and Transplantation in the US- Statistics and Procedures Moderated Debate: Living Organ Donation: Halal or Haram? Facilitated Group Discussions with Peer Educators
  Other Names: Experimental
Other: End of Life Care Workshop — Discussion Moderated by Peer Educators Didactic Session 1: Critical Theological Concepts about Sickness and Health in Islamic Bioethics Didactic Session 2: Islamic Rulings about Brain Death, and Withdrawing/Withholding Life Support Moderated Panel Discussion: End-of-life Decision Making Facilitated Group Discussions with Peer Educators
  Other Names: Control

SUMMARY:
The purpose of this projects is to test the effectiveness of a tailored educational intervention in increasing knowledge about organ donation among Muslim Americans. More specifically, using the theory of planned behavior (TPB) as a conceptual framework, the workshop's goal is to enhance attendee knowledge of the benefits and risks (behavioral beliefs and attitude), understanding of religious arguments for and against (normative beliefs and subjective norm), and procedural knowledge about the process and types of (control beliefs and perceived control) living organ donation.

DETAILED DESCRIPTION:
The study consists of two workshops (control and experimental) and an optional follow-up interview.

The study contains 2 intervention arms based on the order in which the organ donation workshop is delivered at the mosque: early and late. The early arm will receive the experimental organ donation workshop first, followed by the control workshop (on end-of-life care). The late arm will receive the workshops in the opposite order (end-of-life care workshop followed by the organ donation workshop).

To address varied adult learning styles, the workshops will incorporate didactic teaching, moderated panel presentations, and facilitated small group discussions led by a trained peer educator. Workshops will also involve self-administered surveys.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified Muslim men and women
* Fluent in English
* Adult
* Availability to attend workshop sessions

Exclusion Criteria:

* No personal or immediate family history of organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-08-03 (Actual); Study Completion 2019-08-03 (Actual)

PRIMARY OUTCOMES:
Change in Islamic knowledge of living organ donation | 2 weeks
  Islamic Knowledge of Living Donation [IK-LOD] Scale
Change in living organ donation knowledge | 2 weeks
  Living Donation subscale of the Rotterdam Renal Transplant Knowledge Test (R3K-T)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Quinn, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Padela AI, Duivenbode R, Saunders MR, Quinn M, Koh E. The impact of religiously tailored and ethically balanced education on intention for living organ donation among Muslim Americans. Clin Transplant. 2020 Dec;34(12):e14111. doi: 10.1111/ctr.14111. Epub 2020 Nov 1. PMID 33063912
- [Derived] Padela AI, Duivenbode R, Quinn M, Saunders MR. Informing American Muslims about living donation through tailored health education: A randomized controlled crossover trial evaluating increase in biomedical and religious knowledge. Am J Transplant. 2021 Mar;21(3):1227-1237. doi: 10.1111/ajt.16242. Epub 2020 Sep 15. PMID 32772460